CLINICAL TRIAL: NCT03692143
Title: Effect and Cost Comparation of Different Treatment Strategies for Osteoporotic Vertebral Fractures (OVF): Teriparatide Injection and Percutaneous Vertebroplasty (PVP)
Brief Title: Comparation of Treatment Strategies for OVF: Teriparatide Injection and PVP
Status: Active, not recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2018-067
Record Dates: First submitted 2018-09-19; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis, Postmenopausal; Vertebral Fracture; Quality of Life
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Spinal Fractures | interventions — Teriparatide; Alendronate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- teriparatide group: The group of postmenopausal women who diagnosis with osteoporotic fractures treated with teriparatide
  Interventions: Drug: Teriparatide
- PVP group plus alendronate: The group of postmenopausal women who diagnosis with osteoporotic fractures treated with vertebroplasty. Then alendronate was prescribed.
  Interventions: Procedure: PVP; Drug: Alendronate
- teriparatide and PVP group: The group of postmenopausal women who diagnosis with osteoporotic fractures treated with teriparatide after vertebroplasty
  Interventions: Drug: Teriparatide; Procedure: PVP

INTERVENTIONS:
Drug: Teriparatide — subcutaneous injection of teriparatide(20 mg) once daily
  Groups: teriparatide and PVP group; teriparatide group
Procedure: PVP — With local anesthesia, bone cement was injected in to fractured body in a needle that penetrated transpedically and percutaneously
  Groups: PVP group plus alendronate; teriparatide and PVP group
Drug: Alendronate — Alendronate Sodium, oral, 70mg, once a week
  Groups: PVP group plus alendronate

SUMMARY:
This study aimed to compare teriparatide treatments and PVPs, focusing on its effects on life qualities and effect/coast ratio and evaluate which method is better for patients.

DETAILED DESCRIPTION:
Osteoporosis and osteoporotic vertebral fracture (OVF)s are the common diseases that affect the qualities of senior people. The general treatments for OVFs including percutaneous vertebroplasty (PVP) operation and conservative treatments with pain killers. But with the widely used methods, the life quality of patients were still not satisfied. Teriparatide has been proven to increase bone qualities in patients with severe osteoporosis and reduced the fracture possibilities. The investigators' previous clinical observation found teriparatide could be applied to treat fresh OVFs.

90 participants who diagnosed fresh OVFS were included in the trial. After they received each of three kinds of interventions mentioned in this study, The investigators followed up all these cases. Once 30 cases goal reaches in a certain group, the data collection in that special will stop automatically. The quality of life, pain score and BMDs will be evaluated in certain time during the trial.

ELIGIBILITY:
Inclusion Criteria:

* 1.postmenopausal women with osteoporotic fractures 2.treated with teriparatide 3.or treated with vertebroplasty 4.or treated with teriparatide after vertebroplasty 5.or treated with Fosamax 6. willing to anticipate the trial

Exclusion Criteria:

* Serious other illness or disease which effecting quality of life occurs later in treatment
* unwilling to anticipate the trial

Ages: 49 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: postmenopaual women with osteoporotic vertebral fractures, reveived treatments with teriparatide, PVP, teriparatide after PVP, or fosamax only.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life of the patients | Change from pre treatment at 3 months, 6 months, 1 year and 2 years post treatment
  The quality of life will be evaluated with SF-36 questionaire

SECONDARY OUTCOMES:
Pain cause by the fracture | Change from pre treatment at 3 months, 6 months, 1 year and 2 years post treatment
  VAS score will be used to evaluate the pain caused by OVF
Bone healing | 3 month after treatment
  Bone healing will be evaluated with MRI scanning
Bone mineral density | Change from pre treatment at 6 months, 1 year and 2 years post treatment
  Bone mineral density will be evaluated with DEXA.

CONTACTS AND LOCATIONS:
Overall Officials: Dehong Yang, MD,PhD, Principal Investigator — Nanfang Hospital, Southern Medical University

REFERENCES:
- [Derived] Xie Y, Niu S, Ma Y, Liao Y, Zhu Y, Feng L, Zheng M, Yang D. Sequential anti-osteoporotic therapy with teriparatide and alendronate optimizes outcomes of percutaneous vertebroplasty in acute osteoporotic vertebral fractures: a 12-month prospective cohort study. BMC Musculoskelet Disord. 2025 Oct 29;26(1):1011. doi: 10.1186/s12891-025-09256-w. PMID 41163205